CLINICAL TRIAL: NCT00969631
Title: Combined Metformin and Clomiphene Citrate Versus Laparoscopic Ovarian Diathermy for Ovulation Induction in Clomiphene-resistant Women With Polycystic Ovary Syndrome
Brief Title: Combined Metformin and Clomiphene Citrate (CC) or Laparoscopic Ovarian Diathermy for Women With CC Resistant Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU- 012; FMH-009-C
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; clomiphene resistance; metformin; laparoscopic ovarian diathermy
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin-CC (Experimental)
  Interventions: Drug: metformin HCl (Cidophage®; CID,Cairo, Egypt), CC (Clomid®; Global Napi Pharmaceuticals,Cairo, Egypt),Cairo, Egypt)
- Laparoscopic ovarian diathermy (LOD) (Active Comparator)
  Interventions: Procedure: Laparoscopic ovarian diathermy (LOD)

INTERVENTIONS:
Drug: metformin HCl (Cidophage®; CID,Cairo, Egypt), CC (Clomid®; Global Napi Pharmaceuticals,Cairo, Egypt),Cairo, Egypt) — metformin HCl 1500 daily for 6-8 weeks then 100 mg CC for 5 days starting from day 3 of menstruation up to 6 cycles.
  Arms: Metformin-CC
Procedure: Laparoscopic ovarian diathermy (LOD) — Three-puncture technique. Each ovary was cauterized at four points, each for 4 seconds at 40 W for a depth of 4 mm with a mixed current, using an monopolar electrosurgical needle.
  Arms: Laparoscopic ovarian diathermy (LOD)

SUMMARY:
The purpose of this study is to compare and determine the efficacy of combined metformin and Clomiphene citrate administration to that of laparoscopic ovarian diathermy (LOD) in infertile women with Polycystic ovary syndrome (PCOS) not responding to treatment with Clomiphene alone.

DETAILED DESCRIPTION:
All patients in the combined metformin-CC group received metformin HCl (Cidophage®;Chemical Industries Development,Cairo, Egypt), 500 mg thrice daily for 6-8 weeks. Then after the end of this period, they received 100 mg CC (Clomid®; Global Napi Pharmaceuticals,Cairo, Egypt) for 5 days starting from day 3 of menstruation (increased by 50 mg in the next cycle in case of anovulation ). Patients continued treatment for up to six cycles. Metformin was stopped only when pregnancy was documented. All patients in the control group underwent laparoscopic ovarian diathermy, then followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* CC resistant PCOS

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing syndrome
* Androgen secreting tumors

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 282 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
occurrence of ovulation and midcycle endometrial thickness (mm).

SECONDARY OUTCOMES:
occurrence of pregnancy, miscarriage, multiple pregnancy and live birth rates.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. MRCOG, Principal Investigator — Mansoura University Hospital; Naser El Lakany, MD, Study Director — Mansoura University Hospital; Lotfi Sherief, MD, Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals, OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Siebert TI, Kruger TF, Steyn DW, Nosarka S. Is the addition of metformin efficacious in the treatment of clomiphene citrate-resistant patients with polycystic ovary syndrome? A structured literature review. Fertil Steril. 2006 Nov;86(5):1432-7. doi: 10.1016/j.fertnstert.2006.06.014. Epub 2006 Sep 27. PMID 17007847
- [Background] Bayram N, van Wely M, Kaaijk EM, Bossuyt PM, van der Veen F. Using an electrocautery strategy or recombinant follicle stimulating hormone to induce ovulation in polycystic ovary syndrome: randomised controlled trial. BMJ. 2004 Jan 24;328(7433):192. doi: 10.1136/bmj.328.7433.192. PMID 14739186
- [Background] Farquhar C, Lilford RJ, Marjoribanks J, Vandekerckhove P. Laparoscopic 'drilling' by diathermy or laser for ovulation induction in anovulatory polycystic ovary syndrome. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD001122. doi: 10.1002/14651858.CD001122.pub3. PMID 17636653